CLINICAL TRIAL: NCT04369690
Title: How Are You Coping? Assessing the Psychological, Social, and Economic Impacts of an Emerging Pandemic
Brief Title: The Psychological, Social, and Economic Impacts of COVID-19
Acronym: C19Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Ottawa (Other)
Collaborators: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other); Sunnybrook Health Sciences Centre (Other); Southlake Regional Health Centre (Other); The Ottawa Hospital Research Institute (Unknown); Centre for Addiction and Mental Health (Other); Cheo Research Institute (Other); Ottawa Heart Institute Research Corporation (Other); McGill University (Other); Johns Hopkins University (Other); Université de Montréal (Other); The Royal's Institute of Mental Health Research (Other)
Responsible Party: Principal Investigator, Rébecca Robillard, Dr. Rebecca Robillard, University of Ottawa
Other Study IDs: 2131
Record Dates: First submitted 2020-04-20; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Chronic Disease; Psychiatric Disorder; Cardiovascular Diseases
Keywords: COVID-19; pandemic; psychology; social interactions; financial impacts; mental health; stress; anxiety; depression; healthcare professional's health; familly; sleep; occupational life; survey; social media; access to care; social distancing
MeSH Terms: conditions — COVID-19; Chronic Disease; Mental Disorders; Cardiovascular Diseases; Psychological Well-Being; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A dynamic analytical tool is being implemented to monitor the health, psychosocial and economic impacts of the COVID-19 pandemic as the crisis unfolds. A longitudinal survey is distributed via a network of hospitals, provincial/national organizations and web platforms. The survey information can be linked to provincial health administrative data and metrics derived from social media activity based on artificial intelligence methods. Targeted questions are included for critical populations such as healthcare workers and people with chronic illnesses.

DETAILED DESCRIPTION:
The current situation unfolding with regards to the COVID-19 virus is changing core aspects of people's lives in a unique manner. This study aims to examine the psychological, social, and financial impacts of the COVID-19 pandemic at various stages of the outbreak.

Individuals 12 years and older are recruited from three main groups: general population, people with chronic illnesses and healthcare professionals.

An online survey is distributed via multiple hospitals, provincial/national organizations, and web-based platforms at various phases of the outbreak. The survey includes validated questionnaires and custom-made questions to asses the current situation. It notably addresses the following themes: demographics, COVID-19 symptoms and diagnoses, social distancing practices and social interactions, living situation, financial situation, family and work-related challenges, access to healthcare, as well as sleep, physical and mental health.

The survey is available in English and French. It is built on a decisional tree structure with customized subsets of questions based on previous answers.The survey contains an adolescent version and an adult version, and also includes targeted questions for individuals with a current diagnosis of a mental/medical illness. Consent is also sought to link data from parent-child dyads to enable finer analyses of family dynamics. Healthcare staff are invited to answer questions about work-related difficulties, usefulness of virtual tools for clinical practice, as well as moral distress and moral resilience in the context of clinical practice. Healthcare staff who are short on time can chose fill out an abbreviated version. Participants have the option of enabling linkage to linked to provincial health administrative data, and to provide their twitter and facebook handle for social media and mood monitoring through artificial intelligence algorithms. Participants have the option of being followed longitudinally during and after the outbreak.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who are at least 12 years of age

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from 3 groups: general population, individuals with chronic illnesses, and healthcare professionals
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-03 (Actual); Primary Completion 2021-04-03 (Estimated); Study Completion 2021-04-03 (Estimated)

PRIMARY OUTCOMES:
Mental health - Stress | through study completion, estimated to 8 months
  Cohen's Perceived Stress Scale (scores ranged from 0 to 40, higher scores indicating worse stress)
Mental health - Anxiety | through study completion, estimated to 8 months
  Generalized Anxiety Disorder Scale (scores ranged from 0 to 21, higher scores indicating worse anxiety)
Mental health - Depression | through study completion, estimated to 8 months
  Quick Inventory of Depressive Symptomatology-Self-report, short version (scores ranged from 0 to 27, higher scores indicating worse depression)

SECONDARY OUTCOMES:
Moral distress in healthcare workers | through study completion, estimated to 8 months
  Measure of Moral Distress - Healthcare Professionals (scores ranged from 0 to 432, higher scores indicating worse moral distress)
Moral resilience in healthcare workers | through study completion, estimated to 8 months
  Rushton Moral Resilience Scale (scores ranged from 1 to 4, higher scores indicating more resiliency)
Social life | through study completion, estimated to 8 months
  Frequency of interacting with other people (daily, weekly, monthly, less often than monthly)
COVID-9 symptoms | through study completion, estimated to 8 months
  Fever, Cough, Difficulty breathing or shortness of breath, Tiredness, Aches and pains, Nasal congestion, Runny nose, Sore throat, Diarrhea (Mild Moderate, Severe, N/A)
Adverse health long-term outcome | 5 years before the outbreak and two years after
  Mortality (Yes/No): https://datadictionary.ices.on.ca/Applications/DataDictionary/Default.aspx
Health care utilization - Inpatient | 5 years before the outbreak and two years after
  Hospitalizations (total number): https://datadictionary.ices.on.ca/Applications/DataDictionary/Default.aspx
Health care utilization - ER | 5 years before the outbreak and two years after
  Emergency Department visits (Total number): https://datadictionary.ices.on.ca/Applications/DataDictionary/Default.aspx
Health care utilization - Outpatient | 5 years before the outbreak and two years after
  Outpatient visits: https://datadictionary.ices.on.ca/Applications/DataDictionary/Default.aspx
Sleep | through study completion, estimated to 8 months
  Pittsburgh Sleep Quality Index (scores ranged from 0 to 21, higher scores indicating worse sleep disturbances)

CONTACTS AND LOCATIONS:
Overall Officials: Rébecca Robillard, PhD, Principal Investigator — University of Ottawa
Locations (10):
- Canada (10):
  - Southlake Regional Health Centre, Newmarket, Ontario
  - CHEO Research Institute, Ottawa, Ontario
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - The Centre for Addiction and Mental Health, Ottawa, Ontario
  - The University of Ottawa Heart Institute, Ottawa, Ontario
  - The Royal's Institute of Mental Health Research, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hôpital en santé mentale Rivière-des-Prairies (CIUSSS du Nord-de-l'Île-de-Montréal), Montreal, Quebec
  - McGill University, Montreal, Quebec
  - University of Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Robillard R, Saad M, Edwards J, Solomonova E, Pennestri MH, Daros A, Veissiere SPL, Quilty L, Dion K, Nixon A, Phillips J, Bhatla R, Spilg E, Godbout R, Yazji B, Rushton C, Gifford WA, Gautam M, Boafo A, Swartz R, Kendzerska T. Social, financial and psychological stress during an emerging pandemic: observations from a population survey in the acute phase of COVID-19. BMJ Open. 2020 Dec 12;10(12):e043805. doi: 10.1136/bmjopen-2020-043805. PMID 33310814
- See also: Survey link — https://uottawapsy.az1.qualtrics.com/jfe/form/SV_5mOy05DenjLI2sB